CLINICAL TRIAL: NCT05683821
Title: BREATHE 2 Cluster-randomized Trial of Health System Changes to Increase Reach of Smoking Cessation Treatments
Brief Title: BREATHE 2 Clinic Stop-Smoking Treatment Outreach Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0973; 2P01CA180945-06 (NIH); A534253 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison); Protocol Version 07/11/2022 (Other: UW Madison)
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Quitting Smoking; Smoking Cessation; Smoking, Cigarette
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking | interventions — Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced outreach (Experimental): Quarterly outreach via letter and applicable patient-preferred modalities, including e-mail and/or text messaging, offering both standard person-to-person treatment options (quitline referral, primary care provider referral, cessation counseling and treatment in a randomized clinical trial) and self-guided, remote treatment options (mailed nicotine replacement therapy samples and/or facilitated enrollment in a Smokefree.gov texting program). Patients in clinics assigned to this arm will also have the option to initiate treatment by phone or online. Patients may also receive outreach calls from Tobacco Care Managers offering the person-to-person treatments at their health systems 1-30 days following a visit to a participating clinic.
  Interventions: Behavioral: Text message smoking treatment; Drug: Nicotine replacement therapy sampling; Combination Product: Wisconsin Tobacco QuitLine Referral; Combination Product: Referral to Primary Care Provider; Combination Product: BREATHE 2 Cessation Study; Behavioral: Additional modalities to learn about and request treatment
- Standard outreach (Active Comparator): One mailed letter at study initiation outlining available person-to-person treatment options (quitline referral, primary care provider referral, cessation counseling and treatment in a randomized clinical trial) and how to initiate treatment by phone. Patients may also receive outreach calls from Tobacco Care Managers offering the person-to-person treatments at their health systems 1-30 days following a visit to a participating clinic.
  Interventions: Combination Product: Wisconsin Tobacco QuitLine Referral; Combination Product: Referral to Primary Care Provider; Combination Product: BREATHE 2 Cessation Study

INTERVENTIONS:
Behavioral: Text message smoking treatment — Facilitated enrollment in an NCI-sponsored text messaging program:
  * SmokefreeTXT (if ready to set a quit date in the next 14 days)
  * Practice Quit (if ready to practice quitting 1-5 days but not ready to quit permanently)
  * Daily Challenges (if not ready to quit, but willing to make some changes)
  Arms: Enhanced outreach
Drug: Nicotine replacement therapy sampling — Participants may request:
  * Nicotine patches that release nicotine slowly over 24 hours, in either 7 mg, 14 mg, or 21 mg doses
  * Nicotine gum or lozenges that release medication quickly and can be used every 1-2 hours to prevent and cope with cravings to smoke, in either 2 mg or 4 mg doses
  Other Names: Nicoderm, Nicorette
  Arms: Enhanced outreach
Combination Product: Wisconsin Tobacco QuitLine Referral — Patients will be offered referral to the Wisconsin Tobacco QuitLine that offers phone counseling and nicotine replacement starter kits (2 week supplies) to people ready to quit smoking, in addition to web-based, text messaging, and mailed support, at no cost to Wisconsin residents.
Combination Product: Referral to Primary Care Provider — Patients who want to talk to their Primary Care Providers about quitting smoking will be encouraged to make an appointment with their provider to receive smoking cessation counseling and to discuss pharmacotherapy options.
Combination Product: BREATHE 2 Cessation Study — Patients who are interested in participating in a separate randomized controlled trial of smoking cessation treatment will be invited to learn about and complete an eligibility screening and consent process for the trial. Those who enter the study receive both counseling and pharmacotherapy.
Behavioral: Additional modalities to learn about and request treatment — Participants in Enhanced Outreach arm clinics will have the option to request e-mail and/or text message communication regarding their smoking treatment options, and to initiate treatment via phone or online survey.
  Arms: Enhanced outreach

SUMMARY:
The purpose of this research study is to see if offering adult primary care patients who smoke combustible cigarettes more frequent outreach, more choices about how they receive that outreach, and more smoking treatment options will increase the use of smoking treatments and help more people quit smoking, when compared against a standard outreach approach. Only patients at participating adult primary care clinics will be eligible for the study. Five clinic sites will be randomized to an enhanced outreach approach, while another 5 will be randomly assigned to standard smoking treatment outreach. Eligible patients at these clinics will be in this study for up to 18 months.

DETAILED DESCRIPTION:
This 2-arm cluster-randomized clinical trial will compare a standard approach to smoking cessation treatment outreach in adult primary care to an enhanced approach offering more frequent outreach, multiple ways to request treatment, and a broader array of treatment options.

The researchers hypothesize that enhanced outreach comprising quarterly messages offering both standard, person-to-person treatment options (quitline services, care from a primary care provider, phone coaching and medication through a clinical trial) and self-guided treatment options (nicotine replacement therapy sampling (2 week supplies of nicotine replacement therapies and/or enrollment in text-message based cessation support via Smokefree.gov text-message programs) will attract more adult primary care patients who smoke to treatment, and will help more participants achieve abstinence from smoking, as indicated by a change in their smoking status from current to former smoking in their electronic health records. The comparison condition is a standard outreach approach comprising a mailed letter informing participants of person-to-person treatment options (quitline services, care from a primary care provider, and/or phone coaching and medication through a clinical trial).

Up to 12,000 adult participants who receive primary care at 10 participating clinic sites and whose electronic health records suggest they smoke will receive smoking cessation treatment outreach for up to 18 months, unless they opt out of participation. Randomization will occur at the clinic site level rather than at the participant level, and an opt-out approach to recruitment will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 years or older
* Meet criteria for inclusion on a smoking registry (based on current smoking status and/or recent diagnosis of nicotine dependence or treatment of nicotine dependence)
* Being seen in a participating clinic in the past 1-3 years, as documented in the EHR
* Having a valid address
* Not having a language other than English listed as preferred language

Exclusion Criteria:

* Invalid address
* Participant opted out of the study within 18 months of initial outreach letter (or were opted out of the study by a legally authorized representative or an activated power of attorney for health care)
* Participant clarification that they did not meet criteria for the smoking registry at the time of initial outreach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12376 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Smoking treatment initiation within 12 months of enrollment | Up to 12 months
  The proportion of study participants who initiate smoking treatment, as recorded in the electronic health record. Rates of smoking treatment initiation will be compared in the Enhanced Outreach and Standard Outreach arms.

SECONDARY OUTCOMES:
Smoking treatment initiation within 18 months of enrollment | Up to 18 months
  The proportion of study participants who initiate smoking treatment, as recorded in the electronic health record. Rates of smoking treatment initiation will be compared in the Enhanced Outreach and Standard Outreach arms.
Conversion from current smoking to former smoking | 12 and 18 months after study enrollment
  Quitting smoking as indicated by a change in smoking status from current to former smoking, as recorded in the electronic health record.
Cost per quit attempt | Up to 18 months
  Estimated costs per assisted quit attempt initiated will be computed.
Cost per quit | Up to 18 months
  Estimated costs per successful attempt (conversion to former smoking status) will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E McCarthy, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Data for this study will be extracted from electronic health records at health systems participating in this research. These data belong to the health systems and not to the research team. As such, individual participant data will not be available to other researchers until and unless the participating health systems authorize such sharing.

DOCUMENTS (1):
  • Informed Consent Form (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT05683821/ICF_000.pdf